CLINICAL TRIAL: NCT03895606
Title: Application of Machine Learning to Predict Postoperative Acute Kidney Injury in Patients Undergoing Cytoreduction and Hyperthermic Intraperitoneal Chemotherapy Using High-resolution, Time-synchronized Physiological Data From Vital Recorder
Brief Title: Prediction of Kidney Injury After Hyperthermic Intraperitoneal Chemotherapy (HIPEC)* With Machine Learning
Acronym: HIPEC
Status: Completed | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Ji-young Kim, Associate professor, Gangnam Severance Hospital
Other Study IDs: 3-2019-0016
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Acute Kidney Injury; Chemotherapy
MeSH Terms: conditions — Acute Kidney Injury | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIPEC: patients undergoing cytoreductive surgery and hyperthermic intraoperative chemotherapy due to carcinomatosis.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — This study is an observational study collecting perioperative data. There is no intervention regarding this study.

SUMMARY:
Patients undergoing cytoreductive surgery with hyperthermic intraoperative chemotherapy (CRS with HIPEC) are prone to postoperative kidney dysfunction. Previous models predicting kidney injury after CRS with HIPEC did not include intraoperative physiologic data. This study is designed to include not only mean arterial pressure but other parameters such as systolic, diastolic arterial pressure, heart rate, oxygen saturation, body temperature, cardiac index, stroke volume variation and many other physical parameters using a data collection system that can record them every 1-7 seconds. The data will be analyzed using machine learning algorithms.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cytoreductive surgery with hyperthermic intraoperative chemotherapy

Exclusion Criteria:

* patients under 19

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cytoreductive surgery with hyperthermic intraoperative chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
number of patients with postoperative acute kidney injury staged by Kidney Disease: Improving Global Outcomes (KDIGO) | during postoperative day 7
  Stage 1: Increased sCr × 1.5 to 1.9 baseline or ≥ 0.3 mg/dl from baseline or urine output < 0.5 ml/kg/h for 6 to 12 h, Stage 2: Increased sCr × 2.0 to 2.9 baseline or urine output < 0.5 ml/kg/h for 12 h, Stage 3: Increased sCr × 3 baseline or ≥ 4 mg/dl or initiation of RRT, or GFR decrease < 35 ml/min/1.73 m2 for patients < 18 years of age or urine output < 0.3 ml/kg/h for 24 h or anuria for 12 h

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severeance Hospital, Seoul, South Korea